CLINICAL TRIAL: NCT03028779
Title: Implementation of Fast-track Surgery Program for Total Hip and Knee Replacement and the Evaluation of the Risks and Benefits for the Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Pascal André Vendittoli, Orthopedist, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MaisonneuveRH2
Record Dates: First submitted 2016-12-22; First posted 2017-01-23 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Orthopedic Procedure
Keywords: Outpatient,fast-track, arthroplasty, Total knee arthroplasty (TKA), Total hip Arthroplasty (THA)
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fast-track total hip or knee arthroplasty (Experimental): Be able to return patient home on the same day of a total hip or knee surgery.
  Interventions: Procedure: Fast-track Total Hip and knee arthroplasty

INTERVENTIONS:
Procedure: Fast-track Total Hip and knee arthroplasty — To be able to do a total knee or hip arthroplasty and return the patient home in less then 24 hours

SUMMARY:
Implementation of Fast-track surgery for total hip replacement and total knee replacement and evaluation of the risks and benefits for the patients.

DETAILED DESCRIPTION:
The primary goal of the study is to evaluate the risk and the possible implementation of the project of the total knee (TKR) or hip (THR) replacement in a fast track setting. The specifics features of such a study are to introduce intervention modalities and care rapidly to minimize and prevent all known complications associated with THR or TKR.

Following a total hip replacement (THR), the length of stay is usually 1 to 3 days and 3 to 5 days for a total knee replacement (TKR). The investigators have developed a new protocol with intensive care giving the possibility to return home in less than 24 hours and want to evaluate the feasibility and security of such a protocol.

To evaluate the security and feasibility of this protocol the investigators want to recruit 150 participants who will agree to enroll in this study.The investigators will evaluate these variables; number of complications occuring within the 12 months fallowing the surgery, number of readmission post-surgery, pain control efficiency, number of blood transfusion needed, length of wound spread, patient satisfaction and the cost of the program implementation. The investigators want to identify the success and failure factors to optimise the program afterwards.

In order to achieve the evaluation, the investigators will compare the data obtain from the 150 patients to the data retrieved in the medical files of the patients that already had the same usual intervention in the past, with the standard length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Patient understanding the conditions of the study and ready to participate for the duration of the study
2. Patient able to give their informed consent
3. Aged between 18 and 75 years
4. Patient needing a primary total hip or knee replacement (not associated with unusual treatment such as bone graft, osteotomy, revision implant, etc.
5. The patient as a family member or a companion available the day of the pre-op evaluation, the day of surgery and at home after the surgery for a week fallowing the surgery
6. Women in age to procreate have to accept to add another contraception method one month fallowing the intake of Emend/ Aprepitant received pre-surgery.

Exclusion Criteria:

1. Living further than 50 Km from Maisonneuve-Rosemont Hospital
2. Lack of services offered by the CLSC (home health care services) in their area
3. BMI over 40
4. Psychiatric desease limiting the participation in the study
5. Pregnancy
6. The need of long therm urinary foley post-op
7. Allergies to sulfinamide or to the other medications intended in the protocol
8. Presenting a cognitive impairment or a communication problem preventing the realisation of the protocol
9. The patient has had a pulmonary embolism or veinous thromboembolism in the past year
10. Necessitating a long therm anticoagulation therapy
11. Under corticotherapy or has received a systemic corticotherapy in the past year (unless a positive confirmation of a cortrosyn test done before the surgery)
12. Subject with a systemic involvement(diabetic, cardiac, renal, hematologic, etc.) necessitating special perisurgical care (intensive care unit, multiples transfusions, dialysis, etc.)
13. Inflammatory or tumoral joint disease ( rheumatoid arthritis, lupus, etc.)
14. Subject presenting a coagulation problem increasing their bleeding risk per and post surgery (ie : thrombocytopenia, hemophilia, etc.)
15. Subject presenting a locomotion problem ,other then to the joint to be replaced, enforcing functional limitations keeping them from mobilizing without technical or physical aid
16. Presenting neurological or balance disorder
17. Having a living space incompatible with post-surgery home care
18. Under treatment with a medication substrate or strong inhibitor of CYP3A4
19. Subject with Clcr < 30 ml/min ( Cockcroft-Gault formula)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-09 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 year
  All complications related with the surgery from pre-surgery to 1 year after the surgery:
  -Adverse events classification using (Clavien-Dindo Scale) Complication meaning the number of : blood loss/transfusion, wound infection, pain control, dressing problems, leg discrepancy, falls, unexpected fallow up phone calls to the assistant, hospital readmission after discharge, neurological impairment (example; drop foot), range of motion impairment following surgery.

SECONDARY OUTCOMES:
The cost of the outpatient procedure evaluation for the TKR or THR | 1 year
  Estimation of the surgery costs and post surgery costs will be evaluated (procedure, surgery time, medication, lab test etc...) Costs for the hospital such as the cost for the surgery and their complications Costs outside the hospital such as the medication and the cost associated with the lost of productivity Lost of productivity; Work Productivity and Activity Impairment test (WPAI)
Health outcome before surgery at medical evaluation | before surgery at medical evaluation up to 3 months before surgery
  EQ 5D health questionnaire
Health outcome 6 months after surgery | 6 months after surgery
  EQ 5D health questionnaire
Patient sex | up to 3 month before surgery
  Patient sex; men or women Surgery date: (yyyy/mm/dd) Name of the surgeon Height in meters weight in kg BMI in kg/m2 Health and medical history Physical status score (ASA)
Patient date of birth | up to 3 months before surgery
  Patient date of birth Surgery date: (yyyy/mm/dd) Name of the surgeon Height in meters weight in kg BMI in kg/m2 Health and medical history Physical status score (ASA)
Surgery Date | Day of surgery
  Surgery date (yyyy/mm/dd) Name of the surgeon Height in meters weight in kg BMI in kg/m2 Health and medical history Physical status score (ASA)
Name of surgeon | Day of surgery
  Name of the surgeon
BMI | up to 3 months before surgery
  BMI in kg/m2
Health and medical history | up to 3 months before surgery
  Health and medical history
Physical status score (ASA) | up to 3 months before surgery
  Physical status score (ASA)
Surgery Time | The day of surgery
  Evaluation of the surgery length in minutes
Type of prosthesis | The day of surgery
  The type of prosthesis Total Knee Replacement (TKR) or Total Hip Replacement (THR)
Operated side; left or right leg | The day of surgery, when patient arrives in OR
  The side on which the patient is having the TKR(total knee replacement) or THR (total hip replacement)
Quantity of blood in mL loss during surgery | Day of the surgery after closing of the surgical site
  Quantity in mL of blood loss during surgery, measured after closing the surgical site.
The time the patient arrives on the treatment floor | The day of surgery when the patient arrives on treatment floor
  The time in hours and minutes at which the patient arrives on the treatment floor
Blood loss in dressing before discharge in % | Day of the surgery before discharge from hospital up to 24h after surgery
  Percentage evaluation of the quantity of blood in the dressing, where on the dressing, the type of dressing and the aspect of the dressing.
Time at discharged from the hospital | Day of surgery,at discharge time up to 24h after surgery
  The time in hours and minutes at which the patient leaves the hospital after discharged from hospital care.
Number of failure to discharge | through study completion up to 2 years
  The number of failure to discharge patient according to the discharged criterias
Pain score before surgery (VAS) | Before surgery at the medical evaluation pre surgery
  Pain evaluation using the visual analog scale (VAS) zero to ten
Pain score after surgery in recovery room (VAS) | Day of surgery, after surgery in recovery room, day 0
  Pain evaluation using the visual analog scale (VAS) zero to ten in recovery room, day 0
Pain score after surgery on treatment floor before discharge (VAS) | Day of surgery before discharge
  Pain evaluation using the visual analog scale (VAS) zero to ten
Pain score 1-3 days after surgery (VAS) | 1-3 day after surgery
  Pain evaluation using the visual analog scale (VAS) zero to ten
Pain score 4 to 6 weeks after surgery (VAS) | 4 to 6 weeks after surgery
  Pain evaluation using the visual analog scale (VAS) zero to ten
Pain score 10 to 12 weeks after surgery (VAS) | 10-12 weeks after surgery
  Pain evaluation using the visual analog scale (VAS) zero to ten
Pain score 6 months after surgery (VAS) | 6 months after surgery
  Pain evaluation using the visual analog scale (VAS) zero to ten
Pain score one year after surgery (VAS) | one year after surgery
  Pain evaluation using the visual analog scale (VAS) zero to ten
Level of hemoglobin outcome before surgery | Before surgery at the medical evaluation pre surgery up to 3 months before surgery
  Blood test done by nurse evaluating the level in g/L
Level of hemoglobin outcome after surgery | Day of surgery, when the patient arrives in the recovery room
  Blood test done by nurse evaluating the level on g/L ,when the patient arrives in recovery room.
Level of hemoglobin outcome 3 to 4 days after surgery | 3 to 4 days after surgery
  Blood test done by nurse evaluating the level of hemoglobine on g/L
Presence of post surgery symptoms in recovery room | Day of surgery, when the patient arrives in the recovery room
  Evaluation of the symptoms after surgery such as syncope, dizziness, nausea, vomit, headaches.
Presence of post surgery symptoms on treatment floor | Day of surgery, when patient arrives on treatment floor
  subjective evaluation of the symptoms after surgery such as syncope, dizziness, nausea, vomit, headaches
Presence of post surgery symptoms before discharge | Day of surgery, before discharge up to 24h after srugery
  subjective evaluation of the symptoms after surgery such as syncope, dizziness, nausea, vomit, headaches
Blood pressure outcome before surgery at the medical evaluation pre surgery | before surgery at the medical evaluation pre surgery
  Measure of blood pressure in mmHg Measure of the pulse in bpm Measure of saturation in % Measure of the oral temperature in Celcius
Pulse outcome before surgery at the medical evaluation pre surgery | before surgery at the medical evaluation pre surgery
  Measure of the pulse in bpm
  Measure of the oral temperature in Celcius
Saturation outcome before surgery at the medical evaluation pre surgery | before surgery at the medical evaluation pre surgery
  measure of saturation in % with index finger
Temperature outcome before surgery at the medical evaluation pre surgery | Before surgery at the medical evaluation pre surgery
  Measure of oral temperature in Celsius with thermometer
Blood pressure outcome in recovery room | Day of surgery,when patient arrives in recovery room
  Measure of blood pressure in mmHg Measure of the pulse in bpm Measure of saturation in % Measure of the oral temperature in Celcius
Pulse outcome in recovery room | Day of surgery, when patient arrives in recovery room
  Measure of the pulse in bpm Measure of saturation in % Measure of the oral temperature in Celcius
Saturation outcome in recovery room | Day of surgery, when patient arrives in recovery room
  Measure of saturation in % with index finger
Temperature outcome in recovery room | Day of surgery, when patient arrives in recovery room
  Measure of oral temperature in Celsius with thermometer
Blood pressure outcome before discharge | Day of surgery, before discharge up to 24hours after surgery
  Measure of blood pressure in mmHg Measure of the pulse in bpm Measure of saturation in % Measure of the oral temperature in Celcius
Pulse outcome before discharge | Day of surgery, before discharge up to 24hours after surgery
  Measure of pulse in bpm Measure of the pulse in bpm Measure of saturation in % Measure of the oral temperature in Celcius
Saturation outcome before discharge | Day of surgery, before discharge up to 24hours after surgery
  Measure of saturation in % with index finger
Temperature outcome before discharge | Day of surgery before discharge up to 24hours after surgery
  Measure of the oral temperature in Celsius with thermometer
Blood pressure outcome at home 1 to 2 days after surgery | at home 1 to 2 days after surgery
  Measure of blood pressure in mmHg
Pulse outcome at home 1 to 2 days after surgery | at home 1 to 2 days after surgery
  Measure of the pulse in bpm
Saturation outcome at home 1 to 2 days after surgery | at home 1 to 2 days after surgery
  Measure of saturation in %
Temperature outcome at home 1 to 2 days after surgery | at home 1 to 2 days after surgery
  Measure of the oral temperature in Celsius
Presence of big toe extension of the operated limb in recovery room | Day of surgery, when patient arrives in recovery room
  Neurological assesment myotomes evaluation; extension of the big toe of the operated limb.
Presence of plantarflexion of the operated limb in recovery room | Day of surgery, when patient arrives in recovery room
  Neurological assesment Myotomes evaluation; plantarflexion of the operated limb.
Presence of dorsiflexion of the operated limb in recovery room | Day of surgery, when patient arrives in recovery room
  Neurological assesment, myotomes evaluation; platarflexion of the operated limb
Dermatomes evaluation of the operated lower limb on treatment floor | Day of the surgery, on treatment floor 4-6 hours after surgery
  Dermatomes; all lower limbs L2 to S1-S2 if normal and comparable to other limb.
Functional evaluation outcome SF-36 at the medical evaluation before surgery | Before surgery at medical evaluation up to 3 months before surgery
  SF-36 health score questionnaire
Functional evaluation outcome, health score (SF-36) 6 months after surgery | 6months after surgery
  SF-36 health score questionnaire
Functional evaluation outcome hip disability and osteoarthritis outcome score (HOOS) at medical evaluation before surgery | Before surgery at medical evaluation up to 3 months before surgery
  HOOS; hip disability and osteoarthritis outcome score questionnaire
Functional evaluation outcome HOOS 6 months after surgery | 6 months after surgery
  HOOS; hip disability and osteoarthritis outcome score questionnaire
Functional evaluation outcome, knee disability and osteoarthritis outcome score (KOOS) at medical evaluation before surgery | Before surgery at medical evaluation up to 3 months before surgery
  KOOS; knee disability and osteoarthritis outcome score questionnaire
Functional evaluation outcome KOOS 6 months after surgery | 6 months after surgery
  KOOS; knee disability and osteoarthritis outcome score questionnaire
Range of motion outcome of the knee or hip at medical evaluation | Before surgery at medical evaluation up to 3 months before surgery
  Range of motion (ROM) of the knee or hip in degrees in flexion using a goniometer
Range of motion outcome of the knee or hip on treatment floor | Day of surgery, 4-6 hours after surgery
  Range of motion (ROM) of the knee or hip in degrees in flexion using a goniometer
Range of motion outcome of the knee or hip 3 days after surgery | 3 days after surgery
  Range of motion (ROM) of the knee or hip in degrees in flexion using a goniometer
Range of motion outcome of the knee or hip 4-6 weeks after surgery | 4-6 weeks after surgery
  Range of motion (ROM) of the knee or hip in degrees in flexion using a goniometer
Range of motion outcome of the knee or hip 10-12 weeks after surgery | 10-12 weeks after surgery
  Range of motion (ROM) of the knee or hip in degrees in flexion using a goniometer
Range of motion outcome of the knee or hip 6 months after surgery | 6 months after surgery
  Range of motion (ROM) of the knee or hip in degrees in flexion using a goniometer
Range of motion outcome of the knee or hip 1 year after surgery | 1 year after surgery
  Range of motion (ROM) of the knee or hip in degrees in flexion using a goniometer
Straight leg raise (SLR) outcome after surgery | 3-4 hours after surgery
  Measure of the height of the leg from the bed to the heel in centimeters
Walk outcome before surgery at at medical evaluation | Before surgery at at medical evaluation up to 3 months before surgery
  Timed up and go (TUG) test
Walk outcome 40 meters walk test at medical evaluation | Before surgery at medical evaluation up to 3 months before surgery
  Measure of time on m /s to walk 40 meters
Walk outcome 6 months after surgery | 6 months after surgery
  Timed up and go (TUG) test
Walk outcome 40 meters walk test 6 months after surgery | 6 months after surgery
  Measure of time on m /s to walk 40 meters
Stairs climb outcome day of surgery | Day of surgery before discharge up to 24hours after surgery
  Stair climb test; how much time it takes in seconds to go up and down a flight of stairs.
Stairs climb outcome 6 months after surgery | 6 months after surgery
  Stair climb test; how much time it takes in seconds to go up and down a flight of stairs

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No